CLINICAL TRIAL: NCT03931642
Title: BLINAtumomab After R-CHOP Debulking Therapy for Patients With Richter Transformation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FILOCLL13-BLINART
Record Dates: First submitted 2019-03-29; First posted 2019-04-30 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Richter Syndrome
MeSH Terms: interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-CHOP- blinatumomab (Experimental): Patients will first undergo a prior debulking therapy including 2 cycles of R-CHOP.
  At Day1 (D1) : Rituximab 375 mg/m² Intravenous (IV) + Cyclophosphamide 750 mg/m² IV + Doxorubicin 50 mg/m² IV + Vincristine 1.4 mg/m² IV.
  From D1 to D5 : Prednisone 60 mg/m² Per Os (PO). Patients with CR and no measurable lesion left will not be treated further in the setting of the present trial. All the remaining patients will be continuing and treating on study with a single cycle of blinatumomab induction therapy : Blinatumomab at 9 μg/d IV by continuous vein infusion from day 1-7, 28 μg/d from day 8-14 and 112 μg/d from day 15-56.
  Patients who achieve an objective response after induction are eligible to receive one further optional cycle of blinatumomab consolidation : blinatumomab 9 μg/d IV by continuous vein infusion from day 1-7, 28 μg/d from day 8-14 and 112 μg/day IV from day 15-28.
  Interventions: Drug: RCHOP; Drug: Blinatumomab

INTERVENTIONS:
Drug: RCHOP — D1 : Rituximab 375 mg/m² IV + Cyclophosphamide 750 mg/m² IV + Doxorubicin 50 mg/m² IV + Vincristine 1.4 mg/m² IV.
  From D1 to D5 : Prednisone 60 mg/m² PO.
Drug: Blinatumomab — Blinatumomab by continuous vein infusion

SUMMARY:
Blinatumomab (BLINCYTO) is a bi-specific T-cell engaging (BiTE®) antibody construct that transiently links CD3-positive T cells to CD19-positive B-cells, inducing T-cell activation and subsequent lysis of tumor cells.

The investigators propose to evaluate the efficacy, safety and tolerability of blinatumomab administered after R-CHOP debulking therapy in patients with Richter Syndrome (RS) of diffuse large B-cell lymphoma (DLBCL) histology.

The investigators hypothesize that 8-week blinatumomab induction therapy leads to Complete Response (CR) rate improvement (revised Cheson criteria) from a baseline of 7percent as observed in the prospective study evaluating R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma according to the revised iwCLL criteria19 with biopsy proven transformation to diffuse large B-cell lymphoma, consistent with RS according to the 2016 WHO classification
* Both patients with previously treated or treatment-naïve CLL are eligible
* Age greater than or equal to 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <3
* Patients must meet the following hematologic criteria at screening, unless they have significant bone marrow involvement of either CLL or RS cells confirmed on biopsy: absolute neutrophil count ≥1.0 G/L, platelet count ≥50 G/L independent of transfusion within 7 days of screening
* Subject must have adequate coagulation, renal, and hepatic function at screening
* Adequate left ventricular ejection function (> 50 %)
* Patients who have undergone prior allogeneic hematopoietic stem-cell transplantation (HSCT) are eligible as long as they do not have significant active graft versus host disease and that their transplant day 0 is > 6 months from their first dose of protocol therapy
* Female patients of child bearing potential must have negative pregnancy test and use an effective method of birth control during treatment period and 48h thereafter; Males must use an effective method of birth control during treatment period and 48h thereafter.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with the Hodgkin variant of RS
* Patients with previously treated RS
* History or presence of clinically relevant disorder affecting the central nervous system (CNS)
* Known active DLBCL in the CNS (confirmed by cerebrospinal fluid analysis)
* Steroids treatment (≥ 20 mg for one week) before inclusion
* HSCT within 6 months before inclusion
* Active graft-versus-host disease
* History of other malignancies, except: i) malignancy treated with curative intent and with no recurrence over the last 5 years ii) adequately treated non-melanoma skin cancer without evidence of disease iii) adequately treated carcinoma in situ without evidence of disease
* History of human immunodeficiency virus
* Hepatitis B or C seropositivity (unless clearly due to vaccination)
* Pregnant or breastfeeding women
* Unwilling or unable to participate in all required study evaluations and procedures.
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form and authorization to use protected health information (in accordance with national and local subject privacy regulations)
* Abnormal screening laboratory values as defined as following: a) serum glutamate oxaloacetate transaminase and/or serum glutamate pyruvate transaminase and/or alkaline phosphatase > or =5 x upper limit of normal (ULN); b) Total bilirubin > or = 1.5 x ULN, unless due to Gilbert's disease; c) Creatinine > or = 2.0 x ULN or creatinine clearance <50 mL/min (calculated).
* Fertile male and female patients who cannot or do not wish to use an effective method of contraception during treatment and for 48h after the final treatment used for the purposes of the study
* Treatment with other investigational agent or participating to another trial within 30 days prior to entering the study
* No affiliated to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Complete remission (CR) rate according to the revised Lugano criteria | at week 16 from baseline
  the objective response rate to one 8-week cycle of blinatumomab following a debulking therapy with 2 R-CHOP cycles

SECONDARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed by CTCAE v4.0 | From the first treatment administration and during treatment period (R-CHOP and blinatomomab)
  safety and toxicity of blinatumomab after 2 cycles of R-CHOP
overall response | At week 16 from baseline, after blinatumomab induction and at week 24 after blinatumomab consolidation.
  Overall response rate (revised Lugano criteria) after the first and second cycle of blinatumomab,
CR rate | After blinatumomab consolidation (total of 4 weeks) at week 24 from the beginning of study treatment.
  CR rate (revised Lugano criteria) after the second cycle of blinatumomab

CONTACTS AND LOCATIONS:
Overall Officials: Romain GUIEZE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (28):
- France (28):
  - Chu Amiens, Amiens
  - CHU ANGERS - Maladies du sang, Angers
  - Ch Cote Basque, Bayonne
  - Hopital Jean Minjoz, Besançon
  - CH de Béziers - Hématologie, Béziers
  - Hôpital Avicenne - Centre de Recherche Clinique, Bobigny
  - CHU Caen - IHBN - Hématologie Clinique, Caen
  - CHU Estaing - Hématologie Clinique Adulte, Clermont-Ferrand
  - CHU Grenoble - Hématologie, Grenoble
  - Centre Hospitalier du Mans, Le Mans
  - Hôpital Saint Vicent de Paul, Lille
  - Centre Léon Bérard - Hématologie, Lyon
  - Institut Paoli-Calmettes - Hématologie Clinique, Marseille
  - HOPITAL SAINT ELOI - Hematologie, Montpellier
  - Hopital E.Muller, Mulhouse
  - CHU DE NANTES - Hematologie clinique, Nantes
  - Hopital Pitie Salpetriere Service Hematologie Clinique - Pavillon de L'Enfant Et Adolescent, Paris
  - CENTRE HOSPITALIER SAINTJEAN - Hématologie Clinique, Perpignan
  - Bordeaux Pessac, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de la Milétrie - Hématologie et Thérapie Cellulaire, Poitiers
  - Hôpital Robert Debré - Hématologie Clinique, Reims
  - CHU Pontchaillou - Hématologie Clinique BMT-HC, Rennes
  - Centre Henri Becquerel - Service Hématologie Clinique, Rouen
  - Hôpital Hautepierre - Hématologie, Strasbourg
  - IUCT ONCOPOLE - Hématologie, Toulouse
  - Hôpital Bretonneau - Hématologie et Thérapie Cellulaire, Tours
  - Hôpitaux de Brabois - Hématologie Adulte, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No